CLINICAL TRIAL: NCT01586221
Title: A Collaborative Music Therapy/Physical Therapy Intervention to Enhance Well-being and Functional Recovery Post-stroke
Brief Title: Music Therapy/Physical Therapy Intervention to Enhance Well-being and Functional Recovery Post-stroke
Acronym: MT/PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-02284
Record Dates: First submitted 2012-04-09; First posted 2012-04-26 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Stroke With Hemiparesis
Keywords: Rehabilitation; Fingers; Grasp; Strength; Brain Function; Physiopathology; Functional Laterality; Psychomotor Performance; Biomechanis; Touch; Music Therapy; Weight-Bearing
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music & Physical Therapy (Other): Subjects will received Music and Physical Therapy in a group setting.
  Interventions: Other: Music & Physical Therapy

INTERVENTIONS:
Other: Music & Physical Therapy — Participants will receive combined Music Therapy and Physical Therapy for 6 Weeks. Two times per week for 1 hour.

SUMMARY:
The purpose of this study is to see if group Music Therapy and Physical Therapy will help in the recovery from stroke. It is hoped that music and physical therapy in a group setting will help physical, mental, and social well-being.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the feasibility and efficacy of an "enriched," combined music therapy/physical therapy (MT/PT) rehabilitation intervention that addresses physical, psychological, and social well-being simultaneously in a group setting to enhance post-stroke recovery. The intervention will be implemented through collaboration between the Nordoff-Robbins Center for Music Therapy at NYU Steinhardt and the Motor Recovery Laboratory at the Rusk Institute of Rehabilitation Medicine, NYU Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write in English
2. Unilateral stroke at least 6 months prior
3. Independent community ambulation with or without assistive devices
4. Presence of at least 5 degrees of active motion in proximal and distal upper extremity joints, suggesting presence of a neural substrate for recovery

Exclusion Criteria:

1. Neurological or psychiatric disease such as clinical depression
2. Hearing deficits
3. History of surgery or other significant injury that could preclude task performance
4. Complicating medical problems such as uncontrolled hypertension, diabetes with signs of neuropathy, and previous neurological illness such as head trauma, prior stroke, epilepsy or demyelinating disease
5. Any factors that may put the subject at significant risk or confound study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Base Line Measurement of Hand Function | Beginning of study
  Participants will be assessed prior to starting therapy:
  - Measurement of current hand motor impairment during a functional grasp and lift tasks

SECONDARY OUTCOMES:
Hand Function after Therapy | After completion of therapy
  Participants will be assessed after 6 weeks of Therapy for:
  * change in hand motor impairment during a functional grasp and lift tasks
  * Hand Function

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Raghavan P, Geller D, Guerrero N, Aluru V, Eimicke JP, Teresi JA, Ogedegbe G, Palumbo A, Turry A. Music Upper Limb Therapy-Integrated: An Enriched Collaborative Approach for Stroke Rehabilitation. Front Hum Neurosci. 2016 Oct 7;10:498. doi: 10.3389/fnhum.2016.00498. eCollection 2016. PMID 27774059